CLINICAL TRIAL: NCT04908501
Title: Health Care Appropriateness Assessment and Support Programme at a University Hospital Centre (CHU) in Bordeaux
Acronym: sPREAdPerti
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/65
Record Dates: First submitted 2021-05-07; First posted 2021-06-01 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Any Conditions
Keywords: (Health care) appropriateness; (Health care) programme assessment; e-feedbacks
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Services of the non-transversal clinical departments of the Bordeaux University Hospital willing to participate to the programme.
  Interventions: Other: Intervention
- Control group: Services of the non-transversal clinical departments of the Bordeaux University Hospital not willing to participate to the programme.

INTERVENTIONS:
Other: Intervention — The program intervention has three focuses : the prioritization of appropriateness indicators, the automation and visualization of the prioritized indicators, and support for practice analysis groups (PAG) based on e-feedback from automated indicators
  Groups: Intervention group

SUMMARY:
Non-appropriateness of care is a common and serious phenomenon that affects healthcare institutions in France. Appropriateness in health care is about adequacy of any type of health care with patient's needs. Relying on structuring innovative tools, the hospital university centre of Bordeaux is implementing a health care appropriateness assessment and support programme ("sPREAd pertinence").

By using a mixed method, the project's main objective is to evaluate programme effectiveness on the improvement of care appropriateness in hospital university centre of Bordeaux. Other assessments are considering impact on: specific care appropriateness indicators, care related adverse events frequency, organizational climate, and work life satisfaction. The economic impact of this program in terms of induced costs and avoided costs will be evaluated. A qualitative approach will be used to identify the programme transferability conditions with a view to produce an Operational Model for the Implementation of Appropriateness at a Healthcare Institution.

DETAILED DESCRIPTION:
Non-appropriateness of care is a common and serious phenomenon that affects healthcare institutions in France. Appropriateness in health care is about adequacy of any type of health care with patient's needs. It means that a health care is necessary and relevant, given a specific indication, with regard to updated practice recommendations or justifications of experts.

The hospital university centre of Bordeaux is making Health care appropriateness a policy priority. Relying on structuring innovative tools, it is implementing a health care appropriateness assessment and support programme ("sPREAd pertinence"). This programme comprises two parts, one regarding interventional aspects and the other concerning assessments.

sPREAd-Pertinence programme's objectives Project's primary objective is to evaluate programme effectiveness on the improvement of care appropriateness in hospital university centre of Bordeaux.

Project's secondary objectives are :

* to assess impact on specific care appropriateness indicators, care related adverse events frequency, organizational climate and work life satisfaction.
* to evaluate the actual use of GAP.
* to measure the costs of implementing the sPREAD Perti program and to identify the additional costs incurred in comparison with the mobilization and support approach to care appropriateness already existing at the Bordeaux University Hospital;
* to compare the costs of the program with the consequences observed in terms of specific care appropriateness improvement, changes in serious adverse events frequency, organizational work climate and work life satisfaction;
* to estimate, if necessary, in terms of avoided costs, the reduction of serious adverse events frequency.
* to identify, using a qualitative approach:

  * The determinants of programme acceptability and efficiency
  * The appropriation by professionals of the mobilization and support program
  * The impact of the program on professional practices: changes in practices and perceived effectiveness
  * The conditions for programme transferability with a view to producing an Operational Model for the Implementation of Appropriateness at a Healthcare Institution Study design The project is based on a mixed method approach. Study design for the quantitative part is a Stepped-Wedge cluster randomized controlled trial, completed by a control group not receiving the intervention. The clusters are the clinical services of the Bordeaux University Hospital. Up to six volunteer clinical services will be randomly selected to determine the order in which they will start the implementation of the intervention. A control group will be made up of clinical services that meet the inclusion criteria and do not belong to the group of six participating services. The control group will receive the usual support for improving the appropriateness of care.

Qualitative section of the project will analyse the mechanisms of program effectiveness using an exploratory approach based on semi-structured interviews and direct observations of PAG.

Global proportion of patient stays appropriate regarding health cares concerned with feedback indicators available at the start of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Services: services of the non-transversal clinical departments of the Bordeaux University Hospital.
* Health professionals: Medical and paramedical professionals working during the day or night in the participating services for at least one month and at least one day per week.
* Patients: Stays of patients hospitalized at the Bordeaux University Hospital benefiting from care targeted by the automated indicators and made available by the feedback system at the start of the trial.

Exclusion Criteria:

* Services of the transversal and medico-technical departments (Medical Imaging department, Biology and Pathology department, Health Products department, Public Health department and Anesthesia-Intensive care department) and department with specific activity.
* Professionals: planning to be absent during the data collection period.
* Patients: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are 3 study populations in this trial: - Health care professionals : medical and paramedical staffs - Patients - Hospital stays
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Global proportion of patient stays appropriate regarding health cares concerned with feedback indicators available at the start of the trial. | Primary outcome is assessed 14 months after the start of the intervention
  This proportion is calculated by dividing the number of appropriate patient stays for all indicators corresponding to targeted health care by the number of patients who received targeted health care for at least one of the indicators.

SECONDARY OUTCOMES:
Appropriate stays proportion specific to each feedback indicator available at the start of the trial | two months before and fourteen months after applying the programme in the first cluster.
  Appropriate stays proportion specific to each feedback indicator available at the start of the trial is calculated as the number of stays appropriate according to the indicator (numerator) over the number of stays concerned by the indicator (denominator);
Incidence density of serious adverse events | two months before and fourteen months after applying the programme in the first cluster.
  Incidence density of serious adverse events measured by a specific data collection in each service using the questionnaires tested in the two France National Surveys on Adverse Events in Healthcare (ENEIS 1 and ENEIS 2);
Dimension Scores of the Comet questionnaire | two months before and fourteen months after applying the programme in the first cluster.
  Dimension Scores of the Comet ("Contexte Organisationnel et Managérial en Etablissement de santé" / Organizational and Managerial Context in Healthcare Establishments) questionnaire measuring the Organizational Climate (for each dimension, proportion of professionals giving the answers "completely agree" or "agree");
Work life satisfaction | two months before and fourteen months after applying the programme in the first cluster.
  Work life satisfaction score measured by the validated ESVP ("Echelle de Satisfaction globale de Vie Professionnelle" / global professional life satisfaction scale) questionnaire. It consists of 5 items and assesses the overall satisfaction of individuals with their work life. This score is calculated by summing the responses to each of the 5 items. The answers materialize a position on a scale of agreement going from "1" (Not at all in agreement) to "7" (Totally in agreement). The possible range of scores on this scale can thus oscillate from 5 (low satisfaction) to 35 (high satisfaction). The higher the score, the greater the perceived satisfaction with work life.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No